CLINICAL TRIAL: NCT01529983
Title: A Comparison of 1550-nm Fractional Photothermolysis Versus Intense Focused Ultrasound for Treatment of Periorbital Wrinkles: A Pilot, Prospective Randomized Control Trial
Brief Title: Fractional Laser vs. Ultrasound for Periorbital Wrinkles
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU55341
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Wrinkles
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fractional photothermolysis (Experimental): Fractional photothermolysis (FP) for treatment of photo- damaged skin is an FDA-approved method for treating facial rhytids. Fractionated treatment with 1550-nm laser is a safe, nonsurgical method for improvement of periorbital rhytides, photodamage, and scarring
  Interventions: Procedure: Laser treatment; Device: High-intensity focused ultrasound
- High-intensity focused ultrasound (Active Comparator): High-intensity focused ultrasound (HIFUS) is an FDA-approved method for periorbital treatment and nonablative tissue tightening. Ultrasound waves induce a vibration in the tissue, generating heat and increasing the tissue temperature within a focal area. The tissue changes depend on amount of heat and exposure duration. These findings are similar to the thermally induced changes within the skin after CO2 laser fractional ablative treatments.
  Interventions: Procedure: Laser treatment; Device: High-intensity focused ultrasound

INTERVENTIONS:
Procedure: Laser treatment — The treated sites are both lower eyelids and lateral orbits. Each side will be randomized to receive 1550nm-fractionated laser treatment on one side and the contralateral side will receive micro-focused ultrasound treatment every 6-8 weeks for a total of 2 treatments
Device: High-intensity focused ultrasound — High-intensity focused ultrasound (HIFUS) is an FDA-approved method for periorbital treatment and nonablative tissue tightening. Ultrasound waves induce a vibration in the tissue, generating heat and increasing the tissue temperature within a focal area. The tissue changes depend on amount of heat and exposure duration. These findings are similar to the thermally induced changes within the skin after CO2 laser fractional ablative treatments.

SUMMARY:
The primary objective of this study is to compare the efficacy of intense focused ultrasound and carbon dioxide-fractionated laser for treatment of periorbital wrinkles.

DETAILED DESCRIPTION:
This is a prospective randomized comparison study comparing the efficacy of micro-focused ultrasound versus fractionated carbon dioxide laser for treatment of periorbital wrinkles. Subjects who meet inclusion and exclusion criteria will be enrolled in the study. The treated sites are both lower eyelids and lateral orbits. Each side will be randomized to receive 1550nm-fractionated laser treatment on one side and the contralateral side will receive micro-focused ultrasound treatment every 6-8 weeks for a total of 2 treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-60 years old male and female subjects with moderate lower eyelid rhytids and crowsfeet
2. Subjects with Fitzpatrick skin type I-III.
3. Subjects who are willing, have the ability to understand and provide informed consent, and are able to communicate with the investigator.

Exclusion Criteria:

1. Subjects who have received injectable soft-tissue augmentation materials to the face, or facial ablative resurfacing, within the past 6 months.
2. Subjects who were received injectable botulinum toxin to the face, or any nonablative laser treatment to the face, within the past 3 months.
3. Subjects who have local infections, open facial wounds, or other significant local skin disease that would interfere with periorbital treatment with energy devices.
4. Subjects who are allergic to lidocaine or prilocaine.
5. Subjects who have a history of abnormal scarring in the treatment area.
6. Subject who have ectropion or or other eyelid disfigurement.
7. Subjects who have history of isotretinoin use in the preceding year
8. Pregnant or lactating individuals

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Global Improvement Scale | 3 months
  Global improvement scale score, as a percent improvement from baseline to 1 and 3 months, respectively, after treatment. Two non-treating dermatologists will independently blindly evaluate the photographs at baseline, 1 and 3 months after treatment; differences will be resolved via a forced agreement process.
Quantitative eyelid laxity scale | 3 months
  Two non-treating dermatologists will independently blindly evaluate the photographs at baseline, 1 and 3 months after treatment; differences will be resolved via a forced agreement process.

SECONDARY OUTCOMES:
Subject Satisfaction | 10 years
  Subject satisfaction will be determined by a satisfaction questionnaire, and subjects will be asked to select the treatment side they preferred
Adverse events | 10 years
  Any adverse events related to the use of the fractionated laser and ultrasound-tightening device (e.g. infection, prolonged erythema, prolonged edema, bleeding, ulceration, erosion or pigmentation) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States